CLINICAL TRIAL: NCT01203293
Title: CBT for Latinos With Generalized Anxiety Disorder in the General Medical Sector
Brief Title: Cognitive Behavioral Therapy (CBT) for Latinos With Generalized Anxiety Disorder in the General Medical Sector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mildred Vera, Professor, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5SC1MH90599-2; 5SC1MH090599 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-09-16 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental)
  Interventions: Behavioral: Cognitive behavior based therapy
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive behavior based therapy — 15-20 individual psychotherapy sessions
  Arms: Cognitive Behavior Therapy
Behavioral: Treatment as usual — Treatment as usual is an active comparator group in which patients are provided referrals to specialty mental health care services or can use any primary or specialty care services available to them in usual care.
  Arms: Treatment as usual

SUMMARY:
The purpose of this project is to implement culturally adapted Cognitive Behavioral Therapy (CBT) based interventions in general health settings that are delivered to reduce Generalized Anxiety Disorder (GAD) symptoms, increase levels of functioning, and improve health-related quality of life.

DETAILED DESCRIPTION:
This project seeks to lay the foundation for an effectiveness trial that will lead to the advancement of CBT based treatments for GAD among Spanish-speaking Latinos, particularly Puerto Ricans. This area of research is important in light of the limited treatment options currently available for Spanish-speakers with GAD and the long-term negative consequences of this condition. Participants in this study are recruited in general health settings. Patients meeting criteria for enrollment will be randomly assigned to receive either cognitive behavior based therapy or treatment as usual. Assessments for all participants will be collected at baseline, post-treatment, and at two months follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GAD
* 18 to 65 years
* Spanish speaker
* able to read and write
* plan to continue receiving services in the health care setting during the next six months

Exclusion Criteria:

* severe cognitive impairment, psychoses, history of bipolar disease, alcohol or drug abuse or dependence
* clinically judged to have a high acute suicide risk
* life-threatening medical condition
* currently receiving psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire | Baseline
Penn State Worry Questionnaire | Week 20
Penn State Worry Questionnaire | Week 28.

SECONDARY OUTCOMES:
SF-36 Social Functioning Scale | Baseline
SF-36 Social Functioning Scale | Week 20
SF-36 Social Functioning Scale | Week 28
Quality of Life Inventory | Baseline
Quality of Life Inventory | Week 20
Quality of Life Inventory | Week 28

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico